CLINICAL TRIAL: NCT04917887
Title: A Prospective, Observational, Long-Term Follow-Up (LTFU) Study to Evaluate the Long-Term Safety of the Krystal Biotech, Inc. Gene Therapy Backbone Products Using HSV-1 Backbone
Brief Title: Long-Term Follow-up Protocol
Status: Recruiting | Type: Observational
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KRYS-LTFU-01
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Dominant Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this prospective, observational, long-term follow-up (LTFU) study is to evaluate the long-term safety profile of the gene therapy products evaluated by Krystal Biotech, Inc. which have a shared backbone of HSV-1, in participants who received at least one dose of investigational product (IP).

DETAILED DESCRIPTION:
Due to the guidelines for gene therapy for vectors which may undergo latency/ reactivation, Krystal Biotech, Inc. has established a Long-Term Follow-up Protocol which will identify and mitigate the long-term risks to the participants receiving their gene therapy products and capture delayed adverse events in participants, annually, for 5-years following the last study visit. Additionally, it will allow the Sponsor to further understand the persistence of the gene therapy products used in their parent treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* All adult and pediatric participants who received at least one gene therapy treatment in a previous Krystal Biotech, Inc. sponsored study, and have discontinued or completed the parent treatment protocol (which do not have the LTFU embedded into the parent protocol), as applicable.
* Consent/Assent must be obtained by the participants (and, parental/legal representative, when applicable) prior to any study-related data being collected.
* Participant is willing and able to adhere to the protocol requirements.

Exclusion Criteria:

* Participants who enroll into a non-Krystal Biotech, Inc. interventional gene therapy clinical trial will be excluded from the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who received at least one treatment of gene therapy from a Krystal Biotech, Inc. sponsored study, will be asked to roll-over to this LTFU protocol upon either premature discontinuation from, or completion of a prior parent treatment protocol. However, if a participant enrolls in a different Sponsor gene therapy trial during the LTFU phase this participant will be dropped out from the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (AE) | 5 years
  Incidence of delayed Adverse Events suspected to be related to a Krystal Biotech HSV-1 vector backbone investigational product.
  A Serious Adverse Event (SAE) is any untoward medical occurrence (whether considered to be related to gene therapy or not) that:
  * Is fatal
  * Is life-threatening (places the participant at immediate risk of death)
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Is a persistent or significant disability/incapacity, or
  * Is a congenital abnormality/birth defect

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Stanford University, Redwood City, California
  - Pediatric Skin Research, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No